CLINICAL TRIAL: NCT03503760
Title: Efficacy of Extremely Low Magnetic Field (ELF) in Fibromyalgic Patients: Effect on Symptoms Severity, Sleep and Quality of Life.
Brief Title: Efficacy of Extremely Low Magnetic Field (ELF) in Fibromyalgic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Alvise Martini, MD, Principal Investigator, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: CESC prot. ELF-925
Record Dates: First submitted 2018-03-20; First posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Fibromyalgia
Keywords: Extremely low magnetic field (ELF); Fibromyalgia impact questionnaire (FIQ); Pittsburgh Sleep Quality Index (PSQI); Short Form-12 of Physical and Mental Health Summary (SF-12); "LIMFA Therapy®" machine from Eywa Srl system
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Patients have been randomized in two groups using "Research randomizer" avaliable at www.randomizer.org.
  The first group of patients "true-sham" received 6 twice a week sessions of true ELF therapy of one hour with "LIMFA Therapy®", following the antinflammatory, analgesic and biorhythm settings of the device. Then, after a wash-out period (three weeks), it received the sham therapy (no therapy) twice a week for three weeks.
  The second group "sham-true" received 6 twice a week sessions of sham therapy (no therapy) and then, after the wash-out period (three weeks), it received 6 session of true ELF therapy twice a week for three weeks.
  A set of questionnaires were administrated: before first session, after first session, after the wash-out period, after second session and after three week follow-up in both groups.
Who Masked: Participant, Care Provider
Masking Description: Participant and care provider were unaware of the treatment as the machine does not make any sound or heat during the session. Only the nurse that physically connect the cable to the generator knows if the patient recieve or not the therapy but she was not involved in clinical evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- true-sham (Experimental): Patients first received the "true" LIMFA Therapy® treatment for 3 weeks followed by 3 weeks of washout and then six "sham" sessions for 3 weeks more.
  Interventions: Device: LIMFA Therapy®
- sham-true (Experimental): Patients first received the "sham" treatment for 3 weeks followed by 3 weeks of washout and then six "true" LIMFA Therapy® sessions for 3 weeks more.
  Interventions: Device: LIMFA Therapy®

INTERVENTIONS:
Device: LIMFA Therapy® — It applies a packages of magneto-electric field sequences having variable geometry, with frequencies and intensities that vary in a range of 0-80 Hertz and 0-100 microTesla, respectively.

SUMMARY:
This is a randomized double-blind crossover study. The investigators applied ELF with a device named "LIMFA Therapy®" to 48 fibromyalgic patients, assigned in two groups (true-sham and sham-true). Fibromyalgia severity was assessed with the Fibromyalgia Impact Questionnaire (FIQ), quality of sleep with the Pittsburgh Sleep Quality Index (PSQI) questionnaire and global quality of life with Short Form-12 of Physical and Mental Health Summary (SF-12) questionnaire.

DETAILED DESCRIPTION:
In the first part of the protocol the group true-sham received 6 twice a week sessions of true ELF therapy of 1 hour, following the antinflammatory, analgesic and biorhythm settings of the device "LIMFA Therapy®". The sham-true group patients received 6 twice a week sessions of sham therapy (no therapy).

During the second part of the protocol, the true-sham group received the sham therapy twice a week for 3 weeks and the sham-true group received the actual true therapy twice a week for 3 weeks.

For the assessment of pain, sleep quality and global quality of life, a set of questionnaires were administrated at specific stages of the protocol. Questionnaires were administrated every three weeks: before the first therapy, after the first course of therapy, after the washout period, after the second course of therapy, and 3 weeks after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients with an established fibromyalgia diagnosis of at least three months according to American College of Rheumatology 2010 modified criteria and no responsive to their current therapy.
* patients were not responsive to amitryptiline, selective serotonin reuptake inhibitor (SSRI) or duloxetine and pregabalin (with a pain reduction below 50% compared to pre-therapy or intolerant to these drugs)
* patients with a pain level measured with Visual Analogue Scale for Pain (VAS) > 50/100.
* patients that had been taking other drugs or food supplements for the treatment of fibromyalgia for at least 6 months.

Exclusion Criteria:

* patients that completed either physiotherapy or acupuncture or behavioral treatment in the last 6 months
* patients that were affected by other painful syndromes or potentially painful syndromes other than fibromyalgia.
* pregnant women
* pace-maker carriers
* oncologic patients
* tuberculotic patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
FIQ | 12 weeks
  Fibromyalgia Impact Questionnaire is a comprehensive questionnaire for evaluation of fibromyalgia severity. The scale range is from 0 to100 and higher values are considered worse outcomes. In the severity analysis a FIQ score from 0 to 38 represents a mild condition, from 39 to 58 represents a moderate condition, and from 59 to 100 a severe condition. A reduction of FIQ between 10 and 20% is related to a clinically significative intervention. (Bennett, R. et al.(2009))

SECONDARY OUTCOMES:
PSQI | 12 weeks
  Pittsburgh Sleep Quality Index questionnaire measures the quality of sleep. The scale range is from 0 to 21. Higher scores are related to worse sleep condition and the best cut-off score is 5: starting from it, people are identified as affected by sleep disorders. A significant reduction of sleep impairment after treatment is one of the secondary outcome.
SF-12 | 12 weeks
  Short Form-12 of Physical and Mental Health Summary measures global quality of life.
  The results consist of two index: Physical Component Summary(PCS) and Mental Component Summary(MCS). The lower outcomes represent a worse physical and mental condition. A significant improvement of quality of life after treatment is one of the secondary outcome.

REFERENCES:
- [Background] Borchers AT, Gershwin ME. Fibromyalgia: A Critical and Comprehensive Review. Clin Rev Allergy Immunol. 2015 Oct;49(2):100-51. doi: 10.1007/s12016-015-8509-4. PMID 26445775
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783
- [Background] Curcio G, Tempesta D, Scarlata S, Marzano C, Moroni F, Rossini PM, Ferrara M, De Gennaro L. Validity of the Italian version of the Pittsburgh Sleep Quality Index (PSQI). Neurol Sci. 2013 Apr;34(4):511-9. doi: 10.1007/s10072-012-1085-y. Epub 2012 Apr 13. PMID 22526760
- [Background] Sarzi-Puttini P, Atzeni F, Fiorini T, Panni B, Randisi G, Turiel M, Carrabba M. Validation of an Italian version of the Fibromyalgia Impact Questionnaire (FIQ-I). Clin Exp Rheumatol. 2003 Jul-Aug;21(4):459-64. PMID 12942697
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Paolucci T, Piccinini G, Iosa M, Piermattei C, de Angelis S, Grasso MR, Zangrando F, Saraceni VM. Efficacy of extremely low-frequency magnetic field in fibromyalgia pain: A pilot study. J Rehabil Res Dev. 2016;53(6):1023-1034. doi: 10.1682/JRRD.2015.04.0061. PMID 28475205
- [Background] Quittan M, Schuhfried O, Wiesinger GF, Fialka-Moser V. [Clinical effectiveness of magnetic field therapy--a review of the literature]. Acta Med Austriaca. 2000;27(3):61-8. doi: 10.1046/j.1563-2571.2000.270210.x. German. PMID 10897384
- [Background] Bennett RM, Bushmakin AG, Cappelleri JC, Zlateva G, Sadosky AB. Minimal clinically important difference in the fibromyalgia impact questionnaire. J Rheumatol. 2009 Jun;36(6):1304-11. doi: 10.3899/jrheum.081090. Epub 2009 Apr 15. PMID 19369473